CLINICAL TRIAL: NCT02132091
Title: The Effect of Intermittent Fasting on Adaptive Oxidative Stress Response and Mitochondrial Biogenesis
Brief Title: Practicality of Intermittent Fasting and Its Effect on Markers of Aging and Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB772011; TL1TR000066 (NIH); UL1TR000064 (NIH); 1P30AG028740 (NIH)
Record Dates: First submitted 2014-05-05; First posted 2014-05-06 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Aging; Metabolism
Keywords: Sirtuins; Calorie Restriction; Intermittent Fasting; Antioxidant; Aging; Metabolism; Mitochondria; Oxidative Stress
MeSH Terms: conditions — Intermittent Fasting | interventions — Vitamin E; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermittent Fasting (Experimental): Intermittent Fasting
  Interventions: Other: Intermittent Fasting
- Intermittent Fasting + Antioxidants (Experimental): Intermittent Fasting; 400 IU Vitamin E; 1000 mg Vitamin C
  Interventions: Other: Intermittent Fasting; Dietary Supplement: 400 IU Vitamin E; Dietary Supplement: 1000 mg Vitamin C

INTERVENTIONS:
Other: Intermittent Fasting — The intermittent fasting paradigm used in this study will require participants to alternate between days of feasting (175% of normal caloric intake) and fasting ( 25% of normal caloric intake). Food will be provided by University of Florida Clinical Research Center with macronutrient composition prepared according to the 2010 Dietary Guidelines for Americans.
Dietary Supplement: 400 IU Vitamin E — once each day in morning; oral pill form
  Arms: Intermittent Fasting + Antioxidants
Dietary Supplement: 1000 mg Vitamin C — 500mg twice each day; morning and evening; oral pill form
  Arms: Intermittent Fasting + Antioxidants

SUMMARY:
Healthy volunteers will be recruited to participate in a ten-week double-blinded crossover trial. The trial will consist of two, three-week periods of intermittent fasting, where subjects receive either antioxidant supplementation or placebo, the ordering of which will be randomly determined. A one-week preconditioning will precede each invention period, and a two week "wash-out" period will follow the first intervention period. Serum-based assays will be performed to assess levels of reactive oxidant species, antioxidant genes, sirtuins, and markers of mitochondrial biogenesis and aging.

The investigators hypothesize that an intermittent fasting diet in healthy young volunteers will improve these markers of cellular aging and that these beneficial effects will be abrogated by the supplementation of antioxidants. This study is a proof-of-principle study that will shed light on the mechanism and effects of IF as an anti-aging dietary intervention in the absence of weight loss. It will inform the design of dietary interventions that are both effective in improving markers of aging and feasible for patients to practice on a long-term basis.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index in the range of 20.0-30.0 kg/m2;
* Age between 19 and 30;
* Stable weight (change <±10%) for 3 months immediately prior to the study
* No history of metabolic disorders (e.g. non-diabetic), cardiovascular disease, or thyroid dysfunction
* No past or present eating disorders
* No acute or chronic inflammatory disorder
* No more than moderate physical activity (i.e.,<3 hour/week of light exercise sessions for the past 3 months)
* No current medications to regulate blood sugar or lipids
* Not donated blood within 56 days of study start date
* No food allergies
* No dietary restrictions (e.g. vegetarianism and vegan)
* No heavy drinking (more than 15 drinks/week)
* No use of tobacco or recreational drugs within past 3 months
* Access to a microwave or stove
* Access to refrigeration

Exclusion Criteria:

* Inflexibility of schedule such that subject cannot attend blood draw appointments
* Unwillingness to pick-up and eat only study-provided food during the 8 weeks in which it is provided and for unwillingness to abstain from travel (>48hrs) during these same 8 weeks of the trial (travel is permitted during wash-out period)
* Unwillingness to abstain from tobacco, alcohol, recreational drugs, resveratrol or antioxidant supplements (other than study-provided) for the duration of study
* Women who are pregnant, breast-feeding or trying to become pregnant

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
SOD2 gene expression (intermittent fasting) | 3 weeks
  Observational outcome examines difference in expression between a normal diet and a 3-week intermittent fasting diet using RNA extracted from venous blood.
  Note: SOD2 = Superoxide-dismutase-2
SOD2 gene expression (antioxidant supplementation) | 3 weeks
  Experimental outcome examining differences between intermittent fasting with supplementation of antioxidants and intermittent fasting alone using RNA extracted from venous blood.
  Note: SOD2 = Superoxide-dismutase-2

SECONDARY OUTCOMES:
GPx1 gene expression (intermittent fasting) | 3 weeks
  Observational outcome examines difference in expression between a normal diet and a 3-week intermittent fasting diet using RNA extracted from venous blood.
  Note: GPx1 = Glutathione peroxidase 1
SIRT1 gene expression (intermittent fasting) | 3 weeks
  Observational outcome examines difference in expression between a normal diet and a 3-week intermittent fasting diet using RNA extracted from venous blood.
  Note SIRT1 = Sirtuin 1
SIRT3 gene expression (intermittent fasting) | 3 weeks
  Observational outcome examines difference in expression between a normal diet and a 3-week intermittent fasting diet using RNA extracted from venous blood.
  Note SIRT3 = Sirtuin 3
mTFA gene expression (intermittent fasting) | 3 weeks
  Observational outcome examines difference in expression between a normal diet and a 3-week intermittent fasting diet using RNA extracted from venous blood.
  Note: mTFA = mitochondrial transcription factor a
NRF1 gene expression (intermittent fasting) | 3 weeks
  Observational outcome examines difference in expression between a normal diet and a 3-week intermittent fasting diet using RNA extracted from venous blood.
  Note NRF1 = Nuclear respiratory factor 1
8oxodG ratio (intermittent fasting) | 3 weeks
  Observational outcome examines difference in expression between a normal diet and a 3-week intermittent fasting diet using DNA extracted from venous blood.
  Note: 8oxodG = 8-oxo-7,8-dihydro-2'-deoxyguanosine/2-deoxyguanosine
8oxoG ratio (intermittent fasting) | 3 weeks
  Observational outcome examines difference in expression between a normal diet and a 3-week intermittent fasting diet using RNA extracted from venous blood.
  Note: 8oxoG ratio = 8-oxo-7,8 dihydroguanosine/guanosine
GPx1 gene expression (antioxidant supplementation) | 3 weeks
  Experimental outcome examining differences between intermittent fasting with supplementation of antioxidants and intermittent fasting alone using RNA extracted from venous blood.
  Note: GPx1 = Glutathione peroxidase 1
SIRT1 gene expression (antioxidant supplementation) | 3 weeks
  Experimental outcome examining differences between intermittent fasting with supplementation of antioxidants and intermittent fasting alone using RNA extracted from venous blood.
  Note SIRT1 = Sirtuin 1
SIRT3 gene expression (antioxidant supplementation) | 3 weeks
  Experimental outcome examining differences between intermittent fasting with supplementation of antioxidants and intermittent fasting alone using RNA extracted from venous blood.
  Note SIRT3 = Sirtuin 3
mFTA gene expression (antioxidant supplementation) | 3 weeks
  Experimental outcome examining differences between intermittent fasting with supplementation of antioxidants and intermittent fasting alone using RNA extracted from venous blood.
  Note: mTFA = mitochondrial transcription factor a
NRF1 gene expression (antioxidant supplementation) | 3 weeks
  Experimental outcome examining differences between intermittent fasting with supplementation of antioxidants and intermittent fasting alone using RNA extracted from venous blood.
  Note NRF1 = Nuclear respiratory factor 1
8oxodG ratio (antioxidant supplementation) | 3 weeks
  Experimental outcome examining differences between intermittent fasting with supplementation of antioxidants and intermittent fasting alone using DNA extracted from venous blood.
  Note: 8oxodG ratio = 8-oxo-7,8-dihydro-2'-deoxyguanosine/2-deoxyguanosine
8oxoG ratio (antioxidant supplementation) | 3 weeks
  Experimental outcome examining differences between intermittent fasting with supplementation of antioxidants and intermittent fasting alone using RNA extracted from venous blood.
  Note: 8oxoG ratio = 8-oxo-7,8 dihydroguanosine/guanosine

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Brantly, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Wegman MP, Guo MH, Bennion DM, Shankar MN, Chrzanowski SM, Goldberg LA, Xu J, Williams TA, Lu X, Hsu SI, Anton SD, Leeuwenburgh C, Brantly ML. Practicality of intermittent fasting in humans and its effect on oxidative stress and genes related to aging and metabolism. Rejuvenation Res. 2015 Apr;18(2):162-72. doi: 10.1089/rej.2014.1624. PMID 25546413